CLINICAL TRIAL: NCT05874414
Title: Phase 1b/2a Study of GNS561 in Combination With Trametinib in Advanced KRAS Mutated Cholangiocarcinoma
Brief Title: Combination of GNS561 and Trametinib in Patients With Advanced KRAS Mutated Cholangiocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GNS561-222-1
Record Dates: First submitted 2023-04-27; First posted 2023-05-24 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-04

CONDITIONS: Cholangiocarcinoma
Keywords: GNS561; Cholangiocarcinoma; Trametinib; Phase1b/2a; Bile Duct cancer
MeSH Terms: conditions — Cholangiocarcinoma; Bile Duct Neoplasms | interventions — trametinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- GNS561+Trametinib (Experimental): Phase 1b Dose Finding Patients will receive GNS561 (50mg QD; 100mg QD; 150mg; 200mg QD) and trametinib (2mg QD; 1.5mg QD; 1mg QD) in a dose escalation/de-escalation design to determine the maximum tolerated dose (MTD) of the combination.
  Experimental:
  Phase 2a Patients will receive GNS561 and trametinib at the recommended dose of the combination determined during Phase 1b
  Interventions: Drug: GNS561 + Trametinib

INTERVENTIONS:
Drug: GNS561 + Trametinib — GNS561: 50mg, 100mg, 150mg, 200mg and trametinib: 1mg, 1.5mg and 2mg
  Other Names: Ezurpimtrostat (GNS561)

SUMMARY:
This is an open-label, multicenter Phase 1b/2a study to evaluate safety, pharmacokinetics (PK), pharmacodynamics (PD) and efficacy of GNS561 in combination with trametinib in Advanced KRAS Mutated Cholangiocarcinoma after failure of standard-of-care first line therapy

ELIGIBILITY:
Inclusion criteria:

1. Histologically confirmed intrahepatic CCA with a documented KRAS mutation.
2. Patients greater than or equal to 18 years of age.
3. Patients must have disease progression that is not amenable to potentially curative treatment.
4. Patients must have received one or two lines of chemotherapy.
5. Patients must have at least one measurable disease by RECIST v1.1.
6. Performance status (ECOG) 0-1.
7. Adequate organ baseline function defined as follows: absolute neutrophil count ≥1000 cells/μL, platelet count ≥75,000 cells/μL, hemoglobin ≥9 g/dL, aspartate aminotransferase or alanine aminotransferase less than or equal to 3 × upper limit of normal, estimated glomerular filtration rate ≥60 mL/min, corrected QT interval by Fridericia's (QTcF) interval ≤470 msec.
8. Women of childbearing potential must present with a negative serum pregnancy test and agree to use adequate contraception during the study and until 6 months after the end of treatment. Male patients with women partners of childbearing potential must agree with the contraception procedures of the study protocol.
9. Patients must be able to understand and be willing to comply with the requirements of the study protocol.
10. Patients participate voluntarily and sign informed consent form(s).

Exclusion criteria:

1. Previous treatment with a MEK inhibitor or autophagy inhibitor.
2. Previous treatment with three or more lines of prior chemotherapy.
3. Extrahepatic CCA with
4. Current evidence of uncontrolled, significant intercurrent illness including, but not limited to, the following conditions:

   1. Cardiovascular disorders: congestive heart failure New York Heart Association ≥ class 2 or left ventricular ejection fraction (LVEF) <50%, arrythmias or cardiac conduction abnormalities. Uncontrolled arterial hypertension or inadequately controlled arterial hypertension, at the discretion of the investigator, based on an average of = >3 BP readings over = >2 sessions.
   2. Patients who have retinal condition (retinal tear, exudate, hemorrhage) or history of retinal vein occlusion or central serous retinopathy or retinal pigment epithelial detachment.
   3. History of interstitial lung disease or pneumonitis.
   4. Patients who have clinically significant pleural effusion or ascites.
   5. Patients who have neurological condition (e.g., tremor, ataxia, hypotension, confusion), history of seizures or active central nervous system metastases.
   6. Impairment of gastrointestinal function or gastrointestinal disease (e.g., diarrhea, active ulcer disease, history of gastrointestinal perforation/hemorrhage, malabsorption or other conditions that under the judgment of the principal investigator (PI) may impair absorption of study drugs).
   7. Patients who are taking antineoplastic drugs for concomitant cancer or history of malignancy other than CCA within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death (e.g., 5-year OS rate > 90%) such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
   8. Any other condition that would, in the Investigator s judgment, contraindicate the patients' participation in the clinical study due to safety concerns or compliance with clinical study procedures (e.g., infection, unable to swallow medication, social/psychological issues, etc).
5. Known active viral hepatitis, including HBV and HCV.
6. Patients with known allergic reaction to quinoline derivatives (e.g., quinine, chloroquine, mefloquine) and/or hypersensitivity to study drugs.
7. Patients who have not recovered for certain AEs due to previous lines of therpay.
8. Female patients who are pregnant or lactating at the time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-08-21 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLT) of GNS561 with trametinib (Phase 1b) | At the end of Cycle 1 (each Cycle is 21 days)
  Defined as Treatment Emergent Adverse Event (TEAE) being at least possibly related to study drug: With Grade ≥ 3 (using NCI CTCAE Version 5.0 or higher as applicable) such as specified in the protocol
Objective response rate (ORR) of the combination of GNS561 with trametinib (Phase 2a) | Up to 11 months (estimated)
  Defined as the proportion of patients with a best overall response of complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)

SECONDARY OUTCOMES:
Duration of response (DoR) | Up to 11 months (estimated)
  Defined as the duration between first documentation of CR or PR to first documentation of disease progression or death using RECIST v1.1
Progression-free survival (PFS) | Up to 11 months (estimated)
  Defined as the time from the date of first dose of study drug to the date of first documented disease progression or death
Time To Progression (TTP) | Up to 11 months (estimated)
  Defined as the time from first dose of study drug to the date of first documented disease progression.
Disease Control Rate (DCR) | Up to 11 months (estimated)
  defined as the proportion of patients with a best overall response of CR or PR or stable disease (SD) using RECIST v1.1
Time To Response (TTR) | Up to 11 months (estimated)
  Defined as the time from first dose of study drug to first documentation of CR or PR using RECIST v1.1
Overall Survival (OS) time | Up to approximately 42 months
  Defined as the time from the date of first dose of study drug to the date of death due to any cause.
Incidence and severity of treatment emergent adverse event (TEAEs), incidence of serious adverse events (SAEs), incidence of TRAEs, incidence of adverse events of special interest (AESIs), rate of treatment discontinuation or interruption for TRAEs | Up to 11 months (estimated)
  graded according to NCI CTCAE v5.0
Incidence of clinically significant changes or abnormalities from physical examinations, ophthalmologic assessments, vital signs, performance scores, laboratory results, ECGs, echocardiograms or multigated acquisition scans | Up to 11 months (estimated)
Drug concentration in plasma for GNS561 and trametinib | Predose to Day 21 of Cycle 1 and predose to Day 21 of Cycle 2 (each Cycle is 21 days)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lichten, M.D., Study Director — Genfit
Locations (11):
- United States (10):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - LA Cancer Network, Los Angeles, California
  - Orlando Health, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University Of Chicago Medical Center, Chicago, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas, MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Comprehensive Cancer Center, Charlottesville, Virginia
  - Froedtert Hospital and the Medical College of Wisconsin, Milwaukee, Wisconsin
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No